CLINICAL TRIAL: NCT04659798
Title: Prospective Non-interventional Study to Investigate the Relationship Between Duration of Treatment (DoT) and Response in Patients With Multiple Myeloma or Systemic AL Amyloidosis Treated in Real-life Clinical Practice
Brief Title: A Study to Investigate the Relationship Between Duration of Treatment and Response in Patients With Multiple Myeloma (MM) or Systemic AL Amyloidosis Treated in Real-life Practice
Acronym: DOrianT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: C16054; U1111-1258-6881 (Registry Identifier: WHO)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with MM: Participants diagnosed with MM who have received treatment within 12 months preceding the enrollment will be observed prospectively. Data will be collected from the participants medical charts and via electronic case report forms (eCRFs).
- Participants with AL Amyloidosis: Participants diagnosed with AL Amyloidosis who have received treatment within 12 months preceding the enrollment will be observed prospectively. Data will be collected from the participants medical charts and via eCRFs.

SUMMARY:
The study will provide information on outcomes in people with multiple myeloma, or systemic AL amyloidosis, or both, under standard care. AL is short for amyloid light-chain. Standard care means the participant will be treated according to their clinic's standard practice. The study sponsor will not be involved in how participants are treated but will provide instructions on how the clinics will record what happens during the study.

The aim of the study is to learn if treatment duration makes a difference in how participants with multiple myeloma or systemic AL amyloidosis respond to their treatment.

During the study, participants will be treated according to their clinic's standard practice. Participants must have started their treatment up to 12 months before taking part in this study. During the study, the participants will visit their clinic every 3 months. These are extra visits to their clinic's standard visits.

DETAILED DESCRIPTION:
This is a prospective non-interventional study to assess the DoT and response in participants with MM or systemic AL amyloidosis in standard clinical practice.

This study will enroll approximately 250 participants (220 with MM and 30 with systemic AL amyloidosis). Participants will be enrolled in 2 groups:

Participants with MM Participants with AL amyloidosis The study will have a prospective data collection of the participants from clinical records and scheduled visits following the routine clinical practice. All participants will receive treatment at study start and this treatment must have been started within 12 months before the participant's enrollment.

This multi-center study will be conducted in Spain. Participants will be followed until 12 months after enrollment. The overall time to participate in this study is approximately 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MM and/or AL amyloidosis according to the IMWG for MM and BSH guidelines for AL amyloidosis.

   MM diagnostic criteria:
   * Smouldering MM- Both criteria must be met:

     1. Serum M protein (Immunoglobulin G [IgG] or IgA greater than or equal to (>=) 30 gram per liter (g/L) or urinary monoclonal protein (M protein) >= 500 milligram per 24 hours (mg/24 h) and/or clonal bone marrow (BM) plasma cells (PCs) 1 percent (%) - 60%.
     2. Absence of myeloma-defining events or amyloidosis.
   * Multiple myeloma- Clonal BM plasma cells >= 10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following myeloma-defining events:

     1. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically:

        * Hypercalcemia: serum calcium greater than (>) 0.25 millimole per liter (mmol/L) (> 1 milligram per deciliter [mg/dL]) higher than the upper limit of normal or >2.75 mmol/L (>11 mg/dL).
        * Renal insufficiency: creatinine clearance (CrCl) less than (<) 40 milliliter per minute (mL/min) or serum creatinine >177 micromole/liter (mcmol/L) (>2 mg/dL).
        * Anemia: haemoglobin (Hb) value of >20 g/L below the lower limit of normal or a Hb value of <100 g/L.
        * Bone lesions: one or more osteolytic lesions on skeletal radiography, computed tomography (CT) or positron emission tomography-computed tomography (PET-CT).
     2. Any one or more of the following biomarkers of malignancy:

        * >=60% clonal BM plasma cells.
        * Involved/uninvolved serum-free light chain ratio >=100.
        * >1 focal lesions on magnetic resonance imaging (MRI) studies (each focal lesion must be >=5 millimeter (mm) in size).

   AL amyloidosis diagnosis:
   * In suspected AL amyloidosis, a histological diagnosis is essential and, where possible, a biopsy should be taken from an apparently affected organ. Alternatively, a subcutaneous abdominal fat aspirate and bone marrow biopsy may be examined for amyloid.
   * Congo red staining with classical apple green birefringence under polarized light should be used to test for the presence of amyloid on any histological specimen.
   * The diagnosis of amyloid requires an experienced laboratory as false negative and false positive diagnoses on the basis of histology are not infrequent. Other (non-AL) amyloid fibril types should be excluded by using immunohistochemistry, deoxyribonucleic acid (DNA) analysis, protein sequencing or mass spectrometry.
2. Under treatment for MM or systemic AL amyloidosis at the time of study entry.
3. Have started treatment up to 12 months before inclusion for MM or systemic AL amyloidosis, irrespective of the treatment regimen.
4. Having first, second, third or fourth line of treatment for MM or systemic AL amyloidosis, irrespective of the treatment regimen.
5. In case of participants with Newly Diagnosed Multiple Myeloma (NDMM) who are candidates to autologous stem cell transplant (ASCT), the ASCT has to be performed before study entry.

Exclusion Criteria:

1. Participants with planned cessation of treatment for MM or systemic AL amyloidosis from participation to the study (example, due to pregnancy).
2. Participating in blinded clinical trials, or in clinical trials with no possibility of obtaining information required in this study, or in clinical trials in which participation in other studies is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with MM or systemic AL amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
DoT | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  DoT is defined as the time between the start of a treatment/regimen and the end of that regimen.
PFS | From date of the initiation of treatment or regimen the participant is receiving at the time of study entry until progression, death, or 1 year after end of treatment (approximately 1 year)
  PFS: time between start of treatment or regimen and progression or death. PFS for MM will be evaluated according to International Myeloma Working Group(IMWG) and defined per European Society for Medical Oncology(ESMO)guideline. Progressive disease(PD)for MM: increase of 25% from lowest confirmed response value in one of the following criteria: Serum M protein(absolute increase must be>=0.5 g/dL; Serum M protein increases >=1g/dL, if the lowest M component was 5g/dL; Urine M protein(absolute increase must be>=200 mg/24h).PFS for AL amyloidosis will be evaluated as per Guidelines of the British Society for Haematology(BSH).PD for AL amyloidosis: progression from complete response(CR)as any detectable M protein or abnormal free light chain(FLC) ratio(involved light chain must double).Progression from partial response(PR)is defined as a 50% increase in serum M protein to>5.0g/L or 50% increase in urine M protein to>200mg/dL(a visible peak must be present)or FLC increase of 50% to>100mg/L.

SECONDARY OUTCOMES:
Time to Next Treatment (TTNT) | From start of current treatment or regimen until start of next treatment or regimen (approximately 1 year)
  TTNT is defined as time between start of current treatment or regimen and start of next treatment or regimen.
Number of Participants Categorized Based on Treatment Regimens Prescribed in Routine Clinical Practice | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  Number of participants will be reported based on treatment regimens prescribed in routine clinical practice including the number of participants based on treatment line (example- first, second, third or fourth line of treatment), the type of regimen (fixed or continuous), the prescribed duration, and the drug combination used. Fixed duration therapy will be defined as regimen prescribed under a fixed number of cycles. Continuous therapy will be defined as a regimen planned to be administered for a prolonged time (example- 2-3 years), without a pre-defined number of cycles, until progression or intolerance of treatment.
Number of Participants Based on Treatment Response Achieved | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  Treatment response as: CR,stringent CR(sCR),very good partial response(VGPR),PR, based on IMWG/ESMO guideline for MM; BSH for AL amyloidosis.For MM;CR:negative immunofixation on serum/urine,disappearance of any soft tissue plasmacytomas,<=5%PCs in BM, sCR:CR/normal FLC ratio,absence of clonal PCs by immunochemistry or 2-4 colour flow cytometry;VGPR:serum/urine M protein level <100 mg/24h,PR:reduction in serum M protein by >=50%and in 24h urinary M protein by >=90%or<200 mg/24h,>=50%decrease in difference between involved/uninvolved FLC levels required in place of M protein criteria, serum-free light assay is also unmeasurable,>= 50%reduction in PCs required in place of M protein provided baseline BM PC percentage was >=30%and >=50%reduction in size of soft tissue plasmacytomas if serum/urine M protein are unmeasurable. For AL amyloidosis;CR:normal FLC levels with normal kappa/lambda ratio, negative serum/urine immunofixations,VGPR:reduction in dFLC to <40 mg/l,PR:50%reduction in dFLC.
Number of Participants Categorized Based on Differences Between Prescribed and Actual DoT, and Reasons for Treatment Discontinuation | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  Participants will be categorized on the basis of difference between prescribed and actual DoT by evaluating treatment duration and reason for treatment discontinuation.
Number of Participants Satisfied With the Treatment | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  Participant satisfaction regarding treatment will be assessed using Treatment Satisfaction Questionnaire for Medication (TSQM) questionnaire V1.4. The TSQM questionnaire, Spanish version, is a generic measure of satisfaction with the prescribed medication consisting of 14 Likert response items of 7 or 5 alternatives, which assess independently: efficacy (3 items), adverse events (AE) (4 items), convenience of treatment (3 items) and overall satisfaction (3 items). Scores range from 0 to 100, with higher score indicates greater satisfaction in that domain.
Number of Participants Categorized Based on Clinical and Sociodemographic Characteristics Influencing the Treatment Prescribed and Satisfaction With Treatment | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
Percentage of Participants With More Than one Neoplasm | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
Percentage of Participants who Achieve the Prescribed DoT According to Treatment Strategy | From start date of treatment reported at study entry until discontinuation of treatment for any reason (approximately 1 year)
  Treatment strategy as fixed duration therapy or continuous therapy. Fixed duration therapy will be defined as regimen prescribed under a fixed number of cycles. Continuous therapy will be defined as a regimen planned to be administered for a prolonged time (example- 2-3 years), without a pre-defined number of cycles, until progression or intolerance of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (14):
- Spain (14):
  - H. Puerta del Mar, Cadiz, Andalusia
  - Hospital Regional Universitario de Malaga (Carlos de Haya), Málaga, Andalusia
  - H. Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - H. Universitario de Araba, Vitoria-Gasteiz, Basque Country
  - C.H.U. Canarias, San Cristóbal de La Laguna, Canary Islands
  - H. Universitario Marques de Valdecilla, Santander, Cantabria
  - H. Universitario de Leon, León, Castille and León
  - C.H. Salamanca, Salamanca, Castille and León
  - H. Universitario Lucus Agusti, Lugo, Galicia
  - C.H.U. Santiago, Santiago de Compostela, Galicia
  - Hospital General Universitario Santa Lucia, Cartagena, Murcia
  - H. Universitario de Cabuenes, Gijón, Principality of Asturias
  - Hospital Universitario de Burgos, Burgos
  - H. Universitario Fundacion Jimenez Diaz, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5ffeb154565ce300294c6ac5